CLINICAL TRIAL: NCT03275051
Title: A Long-term Safety and Efficacy follow-on Study in Participants With Transfusion Dependent Beta-thalassemia Who Have Previously Received OTL-300 (Formerly Know as GSK2696277)) and Completed the TIGET-BTHAL Study
Brief Title: Long-term Follow-up of Subjects Treated With OTL-300 for Transfusion Dependent Beta-thalassemia Study (TIGET-BTHAL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Telethon Institute for Gene Therapy (OSR-TIGET) (Unknown)
Responsible Party: Principal Investigator, Alessandro Aiuti, Dr, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 207757; 2017-001366-14 (EudraCT Number)
Record Dates: First submitted 2017-08-16; First posted 2017-09-07 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Beta Thalassaemia
Keywords: Beta Thalassaemia; previously GSK2696277; Lentiviral vector; TIGET-BTHAL; Gene therapy
MeSH Terms: conditions — beta-Thalassemia | interventions — Safety

STUDY DESIGN:
Intervention Model Description: No study treatment will be administered in this study. Subjects who have received treatment with OTL-300 in and completed study TIGET-BTHAL will be included in this study.
Masking Description: No study treatment will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Subjects who have received treatment with OTL-300 in and completed study TIGET-BTHAL will be included in this study. Subjects received OTL-300 injection administered intraosseously in TIGET-BTHAL study. No study treatment will be administered in this study (207757).
  Interventions: Other: Safety and Efficacy assessments

INTERVENTIONS:
Other: Safety and Efficacy assessments — Safety and efficacy assessment of OTL-300 in subjects with transfusion dependent beta-thalassemia will be performed.

SUMMARY:
OTL-300 is a gene therapy drug product consisting of autologous hematopoietic stem/progenitor cluster of differentiation (CD) 34+ cells genetically modified with a lentiviral vector (GLOBE) encoding the human beta globin gene. The TIGET-BTHAL is a phase I/II study evaluating safety and efficacy of OTL-300 in subjects with transfusion dependent beta-thalassemia for two years post gene-therapy. Subjects with rare disease who have undergone gene therapy are followed for efficacy and possible delayed adverse events. Thus, this study is designed to follow patients who have received gene therapy on TIGET-BTHAL for an additional six years (for a total of eight years).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed study TIGET-BTHAL i.e. who have received treatment and been followed for two years post treatment with OTL-300.
* For adults; capable of giving signed informed consent. For children; informed assent and/or consent in writing signed by the subject and/or parent(s) / legal representative (according to local regulations and age of the subject).

Exclusion Criteria:

* None

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with absence of abnormal clonal proliferation (ACP) | Up to 6 years
  Clonal proliferation describes the selection and reproduction of only one type of cell.
Number of subjects with Polyclonal engraftment | Up to 6 years
  Integration site analysis will be performed on different hematopoietic lineages from peripheral blood and/or bone marrow. Polyclonality of hematopoiesis is defined as >1000 unique integration sites retrieved at specified time points. The number of subjects with polyclonality of hematopoiesis will be estimated.

SECONDARY OUTCOMES:
Number of subjects with reduction in red blood cells (RBC) transfusion volume | Up to 6 years
Number of subjects with reduction in transfusion rate up to transfusion independence | Up to 6 years
Number of subjects with transfusion independence | Up to 6 years
  Transfusion independence is defined as <= 1 transfusion in the previous 6 months.
Hemoglobin (Hb) levels in subjects achieving transfusion independence | Up to 6 years
Number of subjects with sustained engraftment of genetically corrected cells | Up to 6 years
  Engraftment will be assessed by vector-specific quantitative polymerase chain reaction (PCR) on bone marrow. Sustained engraftment is defined as >=0.15 vector copy number (VCN)/genome in bone marrow erythroid cells.
Number of subjects with overall survival | Up to 6 years
  The number of subjects alive over all the trial.
Number of subjects with adverse events (AEs), serious AEs (SAEs) | Up to 6 years
Clinical chemistry laboratory parameters as a measure of safety | Up to 6 years
Hematology laboratory parameters as a measure of safety | Up to 6 years
Urinalysis as a measure of safety | Up to 6 years
Occurrence of viral infections as a measure of safety | Up to 6 years
  Microbiological laboratory tests will be performed to analyze the presence of hepatitis C virus ribonucleic acid (RNA), hepatitis B virus RNA, hepatitis B surface antigen, human T cell lymphotropic virus type 1-2 antibodies. Molecular tests will be performed for human immunodeficiency virus in peripheral blood or plasma.
Screening for occurrence of antibodies against viruses and toxoplasma as a measure of safety | Up to 6 years
  Immunological laboratory tests will be performed to analyze antibodies to Epstein-Barr virus, cytomegalovirus, herpes simplex virus 1-2, varicella zoster virus, toxoplasma.
Functional assessment of cancer therapy-bone marrow transplant (FACT-BMT) scores | Up to 6 years
Short-Form-36 (SF-36) scores | Up to 6 years
  Impact of disease on overall QoL in adults will be measured using the SF-36.
Pediatric Quality of Life (PedsQL) questionnaire scores | Up to 6 years
  The PedsQL 4.0 generic core scale will be used to measure QoL in pediatric subjects.
Evaluation of growth in pediatric subjects | Up to 6 years
  Growth will be assessed by changes in height versus national growth charts and predicted genetic height.
Assessment of hormonal levels in pediatric subjects | Up to 6 years
Changes in puberty status as assessed by clinical examination | Up to 6 years
Changes in puberty status as assessed by Tanner scale (TS) | Up to 6 years
  Puberty will be assessed using TS.
Changes in puberty status as assessed by general questioning | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Orchard Clinical Trials, Principal Investigator — Ospedale San Raffaele- Telething Institute for Gene Therapy (SR-TIGET)
Locations (1):
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy